CLINICAL TRIAL: NCT04841226
Title: Prospective, Multi-Center, Randomized Study to Assess the Ability of the Silq ClearTract™ Urinary Catheter to Reduce Biofilm Formation When Compared to Two Types of Commercially Available Foley Catheters (Silver-Coated Latex and Silicone-coated Latex)
Brief Title: Randomized Study of Silq Urinary Catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Silq Technologies Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STC-001/F
Record Dates: First submitted 2021-04-07; First posted 2021-04-12 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Biofilm Formation; UTI
Keywords: Urinary Catheter; Foley

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Silq ClearTract™ 100% Silicone 2-Way Foley Catheter (Active Comparator): Up to 82 subjects
  Interventions: Device: Long-term indwelling Foley catheter
- Silver-coated Latex 2-Way Foley Catheter (Active Comparator): Up to 82 subjects
  Interventions: Device: Long-term indwelling Foley catheter
- Silicone-coated Latex 2-Way Foley catheter (Active Comparator): Up to 82 subjects
  Interventions: Device: Long-term indwelling Foley catheter

INTERVENTIONS:
Device: Long-term indwelling Foley catheter — Foley Catheter inserted for up to 28-days

SUMMARY:
To assess the ability of the Silq ClearTract™ 100% Silicone 2-Way Foley Catheter to reduce biofilm formation in subjects that require a long-term indwelling Foley catheter when compared to other commercially available urinary catheters.

DETAILED DESCRIPTION:
A prospective, randomized, multi-center, post-market study in subjects that require a long-term indwelling Foley catheter.

A randomly assigned catheter will be inserted using standard techniques. Non-surgical subjects will rate the level of pain associated with the insertion procedure using the visual analog scale (VAS). A urine sample will be collected immediately after catheter insertion, in order to generate a baseline urinalysis and urine culture.

Follow-up visits will be performed on Day 28, or upon catheter removal, whichever occurs first. The catheter will be removed on Day 28 or earlier if clinically indicated. The removed catheter will be processed and sent to the core laboratory for analysis. Urine will be collected immediately prior to catheter removal in order to conduct urinalysis and urine culture. Subject will rate level of pain associated with the removal procedure using the VAS. The subject will also fill out a questionnaire about their experience with the catheterization immediately after catheter removal. Subjects will then be exited from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age ≥ 18 years old;
2. Requiring indwelling 16Fr Foley catheter for at least 7 days;
3. Able and willing to comply with study procedure; and,
4. Able and willing to give informed consent.

Exclusion Criteria:

1. Allergy or sensitivity to any catheter materials used in this study;
2. Known urethral stricture which, in the opinion of the investigator, could influence the subject's evaluation of the catheter;
3. Planned Prophylactic use of antibiotics for CAUTI or any other infection beyond day 1 of the study (catheter implantation);
4. Symptomatic UTI being treated with antibiotics (as determined by the study PI, including at least one of the following: fever, chills, headache, burning sensation, burning of urethra or genital area, blood in urine, foul smelling urine and ≥ 10,000 cfu/mL);
5. Any other infection being treated with antibiotics at the time of catheter implantation;
6. Subjects requiring bladder irrigation during the study (an active voiding trial in surgical subjects prior to catheter removal is allowed);
7. Currently enrolled in another interventional clinical trial;
8. Any other condition that, in the opinion of the investigator, precludes study participation or poses a significant hazard in case of study participation; and
9. Females who are pregnant or breastfeeding or who plan to become pregnant during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2021-12-28 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Biofilm formation | 5 to 7 days
  A core lab will use the BacTiter-Glo Microbial Cell Viability Assay, a well characterized method for quantifying active biomass and biofilm, to determine biofilm formation on explanted catheter samples.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Urology Associates of Southern Arizona, Tucson, Arizona
  - Rancho Los Amigos National Rehabilitation Center, Downey, California
  - West Los Angeles VA Medical Center, Los Angeles, California
  - Tri Valley Urology Medical Group, Murrieta, California
  - Providence Saint John's Health Center, Santa Monica, California
  - The Iowa Clinic, West Des Moines, Iowa
  - Montefiore Medical Center, The Bronx, New York
  - Evergreen Health, Kirkland, Washington